CLINICAL TRIAL: NCT07163130
Title: Transcutaneous Auricular Vagus Nerve Stimulation in Postural Tachycardia Syndrome: a Prospective Cross-over Study
Brief Title: Tragus Stimulation for POTS Treatment
Acronym: TREAT-POTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vassilios Vassilikos, Professor of Cardiology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TREATPOTS3RDCARDIO
Record Dates: First submitted 2025-08-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence: Active - Sham (Other): This arm will undergo active treatment first and then (after a wash-out period) sham treatment.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- Treatment sequence: Sham - Active (Other): This arm will undergo sham treatment first and then (after a wash-out period) active treatment
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation (tVNS) is an emerging therapeutic modality in cardiovascular diseases. tVNS has been shown to exert antiadrenergic and anti-inflammatory effects in humans. Recently, tVNS has been tested in experimental and human POTS, leading to improved autonomic function, reduction of anti-autonomic autoantibodies and inflammatory cytokines.
  Parasym device; Parasym Health, London, United Kingdom Frequency: 20Hz, pulse width: 200μs, amplitude will be individually titrated to 1 mA below the level that caused mild discomfort.

SUMMARY:
Postural Tachycardia Syndrome (POTS) is a form of dysautonomia characterized by an abnormal cardiovascular response to orthostatic challenges. Individuals afflicted with POTS typically exhibit a heart rate increase of more than 30 beats per minute (bpm) within 10 minutes of assuming an upright posture from a supine or sitting position. This abnormal response is often accompanied by symptoms, such as orthostatic intolerance, dizziness, weakness, fatigue, and, in certain instances, syncope. Lately, there is revived interest in POTS, as it has been quite frequently reported as a manifestation of autonomic dysfunction among patients with long COVID. POTS primarily affects the younger demographic, particularly women, and its pathophysiology appears to be multifactorial, involving autonomic neuropathy, hyperadrenergic state, and inadequate blood volume regulation. Diagnostic criteria commonly include a sustained heart rate increase without significant orthostatic hypotension. The pathophysiological mechanisms of POTS are complex and not fully elucidated. Management strategies encompass lifestyle modifications, exercise programs, and pharmacotherapy, but their efficacy is modest.

Transcutaneous auricular vagus nerve stimulation (tVNS) is an emerging therapeutic modality in cardiovascular diseases. tVNS has been shown to exert antiadrenergic and anti-inflammatory effects in humans. Recently, tVNS has been tested in experimental and human POTS, leading to improved autonomic function, reduction of anti-autonomic autoantibodies and inflammatory cytokines. However, the exact patient characteristics that would identify a patient likely to respond to tVNS as well as further mechanistic and clinical endpoints with tVNS have not been explored.

The aim of this study is to assess and characterize in detail the effect of tVNS in patients with POTS. This is a prospective crossover study in patients with POTS. The expected study duration is approximately 15 months from the time the first subject is enrolled to study termination. Patient enrollment is planned to take place at 3-4 major centers in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years
* Diagnosis of POTS, defined as heart rate increase >30 beats/min from supine within 10 minute of standing, in the absence of orthostatic hypotension (>20/10 mm Hg fall in blood pressure), with chronic symptoms (>6 months), and in the absence of other acute causes of orthostatic tachycardia,
* Signed written informed consent by the patient for participation in the study and agreement to comply with the study procedures and the follow-up schedule.

Exclusion Criteria:

* Hypertension (>150 mmHg systolic and >100 mmHg diastolic) based on history or findings at screening.
* Orthostatic hypotension (consistent drop in blood pressure >20/10 mmHg with 10 min of standing)
* History or presence of significant neurological, immunological, or hematological disorders
* Cardiovascular disease, such as myocardial infarction within 6 months
* Patients on renal dialysis.
* Life expectancy of <12 months
* Currently pregnant women or women planning on becoming pregnant ≤ 5 months
* Patients with active implants (such as a cardiac pacemaker, implantable cardioverter-defibrillator, or a cochlear implant)
* Known channelopathy such as Brugada syndrome, long QT syndrome, or Catecholaminergic monomorphic ventricular tachycardia.
* Episodic or permanent complete heart block or 2nd degree atrioventricular block Mobitz 2 or bifascicular block with concurrent 1st degree atrioventricular block
* Congestive heart failure New York Heart Association class IV, defined as shortness of breath at rest, which is refractory to medical treatment (not responding to treatment)
* Inability to comply with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Heart Rate change during the posture test, between the 2 treatment periods (on-treatment versus off-treatment). | Through study completion, up to 16 months from study start date
  Difference in Heart Rate change during the posture test, between the 2 treatment periods (active versus sham). The Heart rate change will be calculated as Standing Heart rate minus Supine Heart rate, the former being defined as the maximal heart rate recorded during a 10-minute period from erection from the supine to the standing position and the latter as the heart rate immediately before standing (the patient will remain at the supine position in a quiet room for at least 5 minutes before rising to the standing position).

SECONDARY OUTCOMES:
Autonomic symptoms assessed using the Malmo POTS Score questionnaire | Through study completion, up to 16 months from study start date

IPD SHARING:
Plan to Share IPD: Undecided